CLINICAL TRIAL: NCT04818749
Title: Combined Intravenous Dexamethasone and Dexmedetomidine as Adjuncts to Popliteal and Saphenous Nerve Blocks in Patients Undergoing Orthopaedic Surgery of the Foot and Ankle. A Randomised, Blinded, Placebo-controlled, Parallel Clinical Trial
Brief Title: Combined Intravenous Dexamethasone and Dexmedetomidine as Adjuncts to Popliteal and Saphenous Nerve Blocks in Patients Undergoing Orthopaedic Surgery of the Foot and Ankle
Acronym: ADJUNCT2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADJUNCT2
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia, Local
Keywords: Regional anesthesia; Dexamethasone; Dexmedetomidine; Adductor canal block; Saphenous nerve block; Popliteal nerve block; Peripheral nerve block
MeSH Terms: interventions — Sodium Chloride; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Randomised, blinded, placebo-controlled, parallel clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial medication will be prepared by unmasked personnel who are not otherwise involved in the trial. The participant, personnel, caregivers, investigators, outcome assessors, and data analysts will be masked to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants allocated to this arm will have placebo administered intravenously before block performance and placebo administered intravenously after induction of general anaesthesia.
  Interventions: Drug: Saline
- Dexamethasone 12 mg (Active Comparator): Participants allocated to this arm will have dexamethasone 12 administered intravenously before block performance and placebo administered intravenously after induction of general anaesthesia.
  Interventions: Drug: Dexamethasone 12 mg
- Dexamethasone 12 mg + dexmedetomidine 1 mcg/kg (Experimental): Participants allocated to this arm will have dexamethasone 12 administered intravenously before block performance and dexmedetomidine 1 mcg/kg administered intravenously after induction of general anaesthesia.
  Interventions: Drug: Dexamethasone 12 mg + dexmedetomidine 1 mcg/kg

INTERVENTIONS:
Drug: Saline — Saline (placebo) will be administered intravenously before block performance and after the induction of general anaesthesia.
  Other Names: Placebo
  Arms: Placebo
Drug: Dexamethasone 12 mg — Dexamethasone 12 mg will be administered intravenously before block performance and saline (placebo) will be administered intravenously after the induction of general anaesthesia.
  Arms: Dexamethasone 12 mg
Drug: Dexamethasone 12 mg + dexmedetomidine 1 mcg/kg — Dexamethasone 12 mg will be administered intravenously before block performance and dexmedetomidine 1 mcg/kg will be administered intravenously after the induction of general anaesthesia.
  Arms: Dexamethasone 12 mg + dexmedetomidine 1 mcg/kg

SUMMARY:
The investigators will investigate the beneficial and harmful effects of combining dexamethasone (12 mg) and dexmedetomidine (1mcg/kg) as adjuncts to popliteal and saphenous nerve blocks in patients undergoing surgery of their foot or ankle.

DETAILED DESCRIPTION:
This is a randomised, blinded, placebo-controlled, multicentre, parallel, 3-arm clinical trial assessing the effects of adjunct intravenous dexamethasone + dexmedetomidine 1mcg/kg versus intravenous dexamethasone 12mg versus intravenous placebo on time to first pain (i.e. block duration) in patients undergoing surgery of the foot or ankle. All participants will receive a sciatic and saphenous nerve block and general anesthesia.

The investigators will randomise participants to either intervention arm. Participants will be allocated according to a computer-generated random allocation sequence with random permuted blocks and stratification by site. The allocation will be concealed in sequentially numbered opaque envelopes that will not be opened before the participant has been allocated to that specific allocation number/envelope. Trained trial personnel not otherwise involved in the trial will prepare the trial medication according to the allocation.

All others involved will be blinded for the entire duration of the trial (participant, carers, investigators, people delivering the intervention, observers/outcome assessors, statisticians). Blinding will not be broken until agreement has been reached within the steering committee regarding the statistical analysis. The trial medication is prepared in identical syringes with 20ml of identically appearing trial medication. The syringes are subsequently marked with 'syringe 1' and 'syringe 2' and delivered to the investigators. Syringe 1 either contains 12mg dexamethasone or saline and will be administered prior to block performance using an infusion pump set to deliver the volume over 12 minutes. Syringe 2 either contains 1 mcg/kg dexmedetomidine or saline and will be administered after block performance and general anesthesia over 30 minutes using an infusion pump, thereby masking the sedative effect of the dexmedetomidine. The investigators will not be present in the operation room during surgery.

The investigators expect little to no attrition bias since the intervention is simple with a short follow-up. The investigators expect some missing data for duration of the motor block, as most participants will have the affected limb immobilized post-surgery, thereby making assessment of return of motor function difficult.

The statistical analysis plan was pre-defined prior to unblinded data becoming available and can be found on: https://doi.org/10.6084/m9.figshare.22491214.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral osseous surgery of the ankle or foot
* General anaesthesia with both a popliteal and a saphenous nerve block for postoperative analgesia
* Age of 18 or above
* American Society of Anaesthesiologists Physical Status Score of 1 to 3
* Body Mass Index of 18 to 40, but a minimum weight of 50 kg.
* For fertile women, negative urine humane choriongonadotropine test and use of safe anti-conception
* Ability to understand the trial protocol, risks, benefits, and provide signed informed consent

Exclusion Criteria:

* Inability to read and understand Danish
* Uncooperativeness (as judged by investigators)
* Participation in another trial involving medication
* Allergy to study medication
* Daily use of opioids above 30 mg/day morphine (or equivalents)
* Daily use of corticosteroids of more than 5 mg prednisolone equivalents within the past one month
* Neurological or musculoskeletal disease making block performance impossible (as judged by investigators)
* Dysregulated diabetes (as judged by investigators)
* Dysregulated anticoagulants (as judged by investigators)
* History of drug or alcohol abuse
* Glaucoma
* Contraindications for paracetamol or opioids
* Contraindications to general anaesthesia
* Other concomitant conditions needing surgery
* Other concomitant traumatic injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Time to first pain (measured in minutes) | 72 hours
  Time to first pain will be recorded by the patient and measured in minutes as the time to first perceived pain in the surgical area. The patient will be asked to record the time and date of their first perceived pain in their trial log. This date and time will be compared to the date and time of block performance as recorded in the electronic Case Report Form. In the event of the patient not experiencing any pain, the time to first pain will be set to 72 hours.

SECONDARY OUTCOMES:
Duration of the motor block (measured in minutes) | 72 hours
  Duration of the motor block will be recorded by the patient and measured in minutes as the time from removal of the needle to the first movement of their calf muscles, and not the first movement of their distal extremity. The patient will record the date and time of their time to first calf muscle movement on the operative side in their trial log. This date and time will be compared to the date and time of block performance as recorded in the electronic Case Report Form. In the event of the patient not regaining movement of their calf muscles, the duration of the motor block will be set to 72 hours.
Quality of sleep (measured on the Numerical Rating Scale) postoperative night 1 | 24 hours
  Quality of sleep will be measured on the Numerical Rating Scale (0 to 10) where '0' points correspond to the worst possible quality of sleep and '10' points correspond to the best possible quality of sleep. The outcome measure will be recorded by the patients in their trial log after the first, second, and third postoperative night.
Quality of sleep (measured on the Numerical Rating Scale) postoperative night 2 | 48 hours
  Quality of sleep will be measured on the Numerical Rating Scale (0 to 10) where '0' points correspond to the worst possible quality of sleep and '10' points correspond to the best possible quality of sleep.
Quality of sleep (measured on the Numerical Rating Scale) postoperative night 3 | 72 hours
  Quality of sleep will be measured on the Numerical Rating Scale (0 to 10) where '0' points correspond to the worst possible quality of sleep and '10' points correspond to the best possible quality of sleep.
Proportion of participants with one or more serious adverse events | 30 days
  Serious adverse events as defined by the ICH-GCP will be collected and reported as the proportion of participants with one or more serious adverse events. Furthermore, the individual serious adverse events will also be reported.
Proportion of participants with one or more adverse events not considered to be serious | 72 hours
  We will record any adverse events not considered to be serious. We will report the proportion of participants with one or more adverse events not considered to be serious and all individual adverse events not considered to be serious.

OTHER OUTCOMES:
Cumulative oxycodone consumption (measured in milligrams) at 24 hours | 24 hours
  Cumulative oxycodone consumption will be recorded in the electronic medical files of the patients during hospitalisation and in their trial log at 24 hours, 48 hours, and 72 hours by the patient after discharge. The patient will be instructed to record whenever they ingest escape oxycodone, as well as record the total amount of ingested escape oxycodone at 72 hours postoperatively. The patient will be instructed to not count in any usual opioid consumption, but only the escape oxycodone provided by the investigators.
Cumulative oxycodone consumption (measured in milligrams) at 48 hours | 48 hours
  Cumulative oxycodone consumption will be recorded in the electronic medical files of the patients during hospitalisation and in their trial log.
Cumulative oxycodone consumption (measured in milligrams) at 72 hours | 72 hours
  Cumulative oxycodone consumption will be recorded in the electronic medical files of the patients during hospitalisation and in their trial log.
Pain (measured on the Numerical Rating Scale) at 24 hours postoperatively | 24 hours
  Pain will be recorded during rest and measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain. The patients will record their perceived pain at 24 hours postoperatively in their trial log.
Average pain (measured on the Numerical Rating Scale) from 0 to 24 hours postoperatively | 24 hours
  Participants will judge their average pain from 0 to 24 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Worst pain (measured on the Numerical Rating Scale) from 0 to 24 hours postoperatively | 24 hours
  Participants will judge their worst pain from 0 to 24 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Pain (measured on the Numerical Rating Scale) at 48 hours postoperatively | 48 hours
  Pain will be recorded during rest and measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain. The patients will record their perceived pain at 48 hours postoperatively in their trial log.
Average pain (measured on the Numerical Rating Scale) from 24 to 48 hours postoperatively | 48 hours
  Participants will judge their average pain from 24 to 48 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Worst pain (measured on the Numerical Rating Scale) from 24 to 48 hours postoperatively | 48 hours
  Participants will judge their worst pain from 24 to 48 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Pain (measured on the Numerical Rating Scale) at 72 hours postoperatively | 72 hours
  Pain will be recorded during rest and measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain. The patients will record their perceived pain at 72 hours postoperatively in their trial log.
Average pain (measured on the Numerical Rating Scale) from 48 to 72 hours postoperatively | 72 hours
  Participants will judge their average pain from 48 to 72 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Worst pain (measured on the Numerical Rating Scale) from 48 to 72 hours postoperatively | 72 hours
  Participants will judge their worst pain from 48 to 72 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Patient satisfaction (added after initiation of the trial, will only be available for a subset of the patients) | 72 hours
  Patients will be inquired about their satisfaction with a peripheral nerve block related to:
  1. Pain during block performance (Numerical Rating Scale (NRS) from 0 to 10).
  2. Discomfort associated with having a blocked extremity (NRS from 0 to 10, 0 no discomfort & 10 worst discomfort).
  3. Pain immediately after block cessation (NRS from '0' to '10').
  4. Overall satisfaction with block (NRS from 0 to 10, 0 worst & 10 best).
  5. If the participant would accept a block in the future (yes/no)
  6. If the participant would recommend a block to others (yes/no).
  7. If the block duration was too long, too short, or adequate.
  8. Satisfaction with content of information regarding block (NRS 0 to 10, 0 worst & 10 best)
  9. Satisfaction with the amount of information regarding block (NRS 0 to 10, 0 worst & 10 best)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Maagaard, MD, Principal Investigator — Department of Anaesthesiology, Zealand University Hospital, Køge, Denmark
Locations (2):
- Denmark (2):
  - Department of Anaesthesiology, Køge, Zealand Region of Denmark
  - Department of Anaesthesiology, Bispebjerg Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data in anonymised form will be shared upon reasonable request to the primary investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When the trial has been completed, data analysed, and trials results published.
Access Criteria: Individual patient data in anonymised form will be shared upon reasonable request to the primary investigator.